CLINICAL TRIAL: NCT05614102
Title: An Open-label, Phase 1, First-in-human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Maximum Tolerated or Administered Dose, Pharmacokinetics, Pharmacodynamics, and Tumor Response Profile of the Diacylglycerol Kinase Zeta Inhibitor (DGKzi) BAY 2965501 as Monotherapy, and in Combination, in Participants With Advanced Solid Tumors
Brief Title: A First-in-human Study to Learn How Safe the Study Drug BAY2965501 is, Find the Best Dose (Single Drug & Combination), How it Affects the Body, What Maximum Amount Can be Given, How it Moves Into, Through and Out of the Body, How it Acts on Different Tumors in Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 21948; 2023-507905-33-00 (Other: EU-CT Number); 2022-002016-23 (EudraCT Number)
Record Dates: First submitted 2022-10-25; First posted 2022-11-14 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Advanced Solid Tumors
Keywords: Solid tumors; Non-small cell lung cancer; NSCLC; Gastroesophageal junction adenocarcinoma; GEJ adenocarcinoma; Renal cell carcinoma; RCC; Melanoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Melanoma | interventions — pembrolizumab; Platinum Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose escalation of BAY2965501 (Experimental): For escalation part, different dose levels of BAY2965501 are planned.
  Interventions: Drug: BAY2965501
- Dose expansion of BAY2965501 (Experimental): For expansion part, specific tumor types are recruited: NSCLC (non-small cell lung cancer).
  Interventions: Drug: BAY2965501
- Dose escalation of BAY2965501+pembrolizumab (Experimental): For escalation part different dose levels of BAY2965501 are planned in combination with 200mg pembrolizumab. BAY2965501 will be taken in combination with 200mg pembrolizumab every 3 weeks.
  Interventions: Drug: Pembrolizumab
- Dose expansion of BAY2965501 +pembrolizumab (Experimental): For expansion part, specific tumor types are recruited (non-small cell lung cancer (NSCLC) and gastric/gastroesophageal junction (GEJ) adenocarcinoma). BAY2965501 will be taken in combination with 200mg pembrolizumab every 3 weeks.
  Interventions: Drug: Pembrolizumab
- Dose escalation of BAY 2965501 + pembrolizumab + platinum-based regimen (Experimental): The starting dose of BAY 2965501 with pembrolizumab for this combination will be no higher than one dose level below that shown to be safe in BAY 2965501 and pembrolizumab dose escalation. The doses of platinum-based regimen will be as per standard of care and given for a maximum of 6 cycles, in line with the current labeled dose. The dose of pembrolizumab will be 200 mg every 3 weeks, in line with the current labeled dose.
  Interventions: Drug: Platinum-based Chemotherapy
- Dose expansion of BAY 2965501 + pembrolizumab + platinum-based regimen (Experimental): Participants with selected (to be decided by the sponsor) advanced solid tumors will be recruited in a dose expansion cohort of BAY 2965501 with pembrolizumab and platinum-based regimen.
  Interventions: Drug: Platinum-based Chemotherapy

INTERVENTIONS:
Drug: BAY2965501 — Daily oral application
  Arms: Dose escalation of BAY2965501; Dose expansion of BAY2965501
Drug: Pembrolizumab — In combination group 200mg as infusion every 3 weeks
  Arms: Dose escalation of BAY2965501+pembrolizumab; Dose expansion of BAY2965501 +pembrolizumab
Drug: Platinum-based Chemotherapy — Standard of care doses per tumor type will be administered.
  Arms: Dose escalation of BAY 2965501 + pembrolizumab + platinum-based regimen; Dose expansion of BAY 2965501 + pembrolizumab + platinum-based regimen

SUMMARY:
Researchers are looking for a better way to treat people who have advanced solid tumors. Advanced solid tumors are types of cancer that may have spread to nearby tissue, lymph nodes, and/or to distant parts of the body and that are unlikely to be cured or controlled with currently available treatments. This study focuses on certain types of skin cancer, kidney cancer, stomach cancer, and lung cancer. The study treatment BAY2965501 is currently under development as monotherapy or in combination for the treatment of people with advanced solid tumors. BAY2965501 blocks an enzyme in T-cells to activate them. T-cells are a type of immune cell that are known to have an anti-cancer effect and BAY2965501 is a potential new immunotherapy. The main purpose of this first-in-human study is to learn: • how safe different doses of BAY2965501 are when given as a single drug or in combination, • the degree to which medical problems caused by BAY2965501 when given as a single drug or in combination, can be tolerated (also called tolerability), • what maximum amount can be given as a single drug or in combination, and • how it moves into, through and out of the body as a single drug or in combination. To answer this, researchers will look at: • the number and severity of medical problems participants have after taking BAY2965501 as a single drug or in combination for each dose level. These medical problems are also referred to as adverse events. • the (average) total level of BAY2965501 in the blood (also called AUC) after intake of single and multiple doses • the (average) highest level of BAY2965501 in the blood (also called Cmax) after intake of single and multiple doses Doctors keep track of all medical problems that participants have during the study, even if they do not think the medical problem might be related to the study treatment. In addition, the researchers want to know if and how the participants' tumors change after taking BAY2965501. The study will have two parts. The first part, called dose escalation, is done to find the most appropriate dose that can be given in the second part. For this, participants will be assigned to receive one of the planned doses and schedules of BAY2965501 as single drug or participants will be assigned to one of the increasing doses of BAY2965501 in combination with 200mg pembrolizumab. Additionally, platinum based chemotherapy as decided by the treating investigator will be given within the first months (at minimum 2 cycles and up to 6 cycles maximum). Here participants will receive BAY 2965501 in combination with pembrolizumab and platinum based chemotherapy.

All participants will take BAY2965501 by mouth. Additionally, in combination group 1, pembrozilumab will be given as infusion using a small tube that goes into your vein. In combination group 2, pembrolizumab and platinum based chemotherapy will be given as infusion using a small tube that goes into your vein.

In the second part, called dose expansion, all participants in the single drug group will receive up to 2 of the most appropriate doses of BAY2965501 from the 1st part as tablet by mouth. The participants in the combination groups (group 1: + pembrozilumab; group 2: + pembrolizumab and platinum based chemotherapy) will receive the most appropriate dose of BAY2965501 from the first part. Participants in both parts of the study, will take the study treatment until the tumor gets worse (also known as 'disease progression'), or until the participants have medical problems. In general, the study treatment is planned for a maximum of 35 cycles. Each participant will be in the study for several months, including a screening phase of up to 28 days, few months of treatment depending on the participant's benefit, and a follow up phase after the end of treatment. Participants in part two will be assigned to one of 3 groups depending on cancer characteristics.During the study, the study team will: • take blood and urine samples • do physical examinations • check vital signs such as blood pressure, heart rate, body temperature • examine heart health using ECG (electrocardiogram) • check if the participants' cancer has grown and/or spread using CT (computed tomography) or MRI (magnetic resonance imaging) and, if needed, bone scan • take tumor samples (if required) The treatment period ends with a visit no later than 7 days after the last BAY2965501 dose in the single drug and combination group. About 30 and 90 days after the last dose and every 12 weeks thereafter, the study team will check the participants' health and any changes in cancer. This follow-up period ends with worsening of the cancer, start of new anti-cancer therapy, or until the participant leaves the study.

ELIGIBILITY:
Inclusion Criteria:

* Have measurable disease per Response evaluation criteria in solid tumors version 1.1 (RECIST 1.1) as assessed by the local site investigator.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Participants with histologically confirmed diagnosis of a solid tumor (specifications for the different parts of the study below) will be enrolled onto this study:

  •Dose escalation (for monotherapy or BAY 2965501 and pembrolizumab combination cohorts): All solid cancers, except primary central nervous system cancers •Dose escalation (for BAY 2965501 with pembrolizumab and platinum-based regimen combination cohorts): All solid cancers, except primary central nervous system cancers, (including Non-small cell lung cancer (NSCLC), head and neck squamous cell cancer (HNSCC), cervical, endometrial, triple negative breast cancer) that are eligible for standard of care platinum-based regimen and for whom this trial is a reasonable option for them.
* The following tumor types may be recruited to the monotherapy expansion cohorts:

  o Non-small cell lung cancer (NSCLC)
* The following tumor types may be recruited to the BAY 2965501 and pembrolizumab combination expansion cohorts:

  * NSCLC: participants who are treatment-naïve in the incurable disease setting.
  * NSCLC: Participants with metastatic NSCLC (confirmed histologically or cytologically)
  * Gastric/GEJ adenocarcinoma
* other tumor types may be explored based on emerging data
* The following tumor types will be recruited to the BAY 2965501 and pembrolizumab with platinum-based regimen combination expansion cohorts:

  * All solid cancers, except primary central nervous system cancers (including NSCLC, HNSCC, cervical, endometrial, triple negative breast cancer), that are eligible for standard of care platinum-based regimen

Exclusion Criteria:

* Previous therapy with a DGK inhibitor other than BAY 2965501 or BAY 2862789 is prohibited. Participants previously treated with BAY 2965501 or BAY 2862789 must have progressed on that DGK inhibitor (given as monotherapy and not have discontinued for toxicity) to be eligible for the combination of BAY 2965501 and pembrolizumab cohorts only.
* Has received a prior therapeutic regimen containing an anti-PD-1, anti-PD-L1, or anti PD-L2 agent or an agent directed to another co-stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137) and was discontinued from that treatment due to a Grade 3 or higher infusion-related adverse event (irAE).
* Participants with new brain metastases on screening brain MRI/CT. Previously treated brain metastases that are progressive at screening compared to a brain MRI/CT at least 4 weeks earlier are also excluded. Participants with known previously treated brain metastases, which are radiologically stable compared to a CT/MRI scan at least 4 weeks earlier, clinically stable and without the requirement of steroid treatment for at least 14 days prior to the first dose of study treatment
* Primary central nervous system malignancy or presence of leptomeningeal disease (i.e., positive cerebrospinal fluid cytology or unequivocal radiological or clinical evidence of leptomeningeal involvement).
* Participants with gastrointestinal conditions that may compromise oral absorption such as short bowel syndrome or active tumor-related bowel obstruction with ongoing symptoms compromising absorption over last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2027-06-07 (Estimated); Study Completion 2027-09-09 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of treatment-emergent adverse events (TEAEs) including treatment-emergent serious adverse events (TESAEs) | Up to 90 days after the last administration of study treatment
Maximum Tolerated Dose (MTD): Number of participants experiencing dose-limiting toxicities (DLTs) at each dose level in the dose escalation part of the study | From first dose of study treatment to the end of Cycle 1 (each cycle is 21 days)
Maximum Administered Dose (MAD): Number of participants experiencing dose-limiting toxicities (DLTs) at each dose level in the dose escalation part of the study | From first dose of study treatment to the end of Cycle 1 (each cycle is 21 days)
Maximum concentration (Cmax) of the respective dosing interval of BAY2965501 after single dose and multiple-dose | From pre-dose up to 24 hours after administration on Cycle 1 Day 1 (each cycle is 21 days)
Area under the curve [AUC (0 - 24)] of the respective dosing interval of BAY 2965501 after single-dose and multiple-dose | From pre-dose up to 24 hours after administration on Cycle 1 Day 1 (each cycle is 21 days)
  If AUC(0-24) cannot be calculated reliably, it might become necessary to appoint the additional parameter AUC(0-tlast) as primary variable.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Approximately 6 months
  Investigator assessment using Response Evaluation Criteria in Solid Tumours version (RECIST 1.1)
Disease control rate (DCR) | Approximately 6 months
  Investigator assessment using Response Evaluation Criteria in Solid Tumours version (RECIST 1.1)
Duration of response (DOR) | Approximately 6 months
  Investigator assessment using Response Evaluation Criteria in Solid Tumours version (RECIST 1.1)
Progression-free survival (PFS) rate at 6 months | At 6 months
  Investigator assessment using Response Evaluation Criteria in Solid Tumours version (RECIST 1.1)
Overall survival (OS) rate at 12 months | At 12 months
Change from baseline in peripheral activation of effector T memory cells as assessed by flow cytometry | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months
Change from baseline in interleukin 2 and interferon-gamma levels after ex-vivo stimulation | Screening, Cycle 1: Day 1, Day 8 (each cycle is 21 days)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (3):
  - Sarah Cannon Research Institute at HCA HealthONE Presbyterian St. Luke's, Denver, Colorado
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - START | San Antonio, San Antonio, Texas
- Belgium (2):
  - Antwerp University Hospital | Oncology Department, Antwerp
  - Ghent University Hospital | Drug Research Unit Department, Ghent
- China (3):
  - Sir Run Run Shaw Hospital, Zhejiang Univ. School of Medicine - Oncology Department, Hangzhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
- National Cancer Center Hospital East, Kashiwa, Chiba, Japan
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggido
  - Severance Hospital, Yonsei University Health System - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (4):
  - Hospital Hm Nou Delfos | Oncologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
  - Clinica Universidad De Navarra | Oncologia, Madrid
  - Hospital Universitario Hm Sanchinarro | Oncologia, Madrid
- United Kingdom (4):
  - Guy's and St Thomas' NHS Foundation Trust - Guy's Hospital, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust | Churchill Hospital - Oncology, Oxford, Oxfordshire
  - Royal Marsden NHS Trust (Surrey), Sutton, Surrey
  - Freeman Hospital, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — https://clinicaltrials.bayer.com/study/21948